CLINICAL TRIAL: NCT03703219
Title: The Role of Indian Post-partum Care in Women's Psychological Functioning
Brief Title: Impact of Mothers Touch Program on Women's Psychological Functioning
Status: Completed | Type: Observational
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Mothers Touch Foundation, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: NMP 0143
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Psychological Distress; Post Partum Depression; Mood
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mother Touch Program: Forty days of rest period of the mother after delivery, Full body massage, diet and belly binding methods were administered by trained carer.
  Interventions: Other: Mothers Touch Program
- Usual care Program: comparison cohort were followed in usual care under the supervision of health professionals.

INTERVENTIONS:
Other: Mothers Touch Program — Combination of diet, massage, body binding methods along with 40 days of rest following the traditional way of delivering
  Groups: Mother Touch Program

SUMMARY:
The study investigates the effect of the Mothers Touch program on the psychological well-being of new mothers following 5 weeks of child birth. Mothers Touch Program is designed based on traditional Indian post-partum care given by trained carer in the family.

Study was designed as cohort, including a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women giving birth for first time (primiparous)
* Given informed consent
* Accepts traditional home care

Exclusion Criteria:

* Previous history of mental health condition
* History drug or substance abuse

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants giving birth in pre selected 4 hospitals in India.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Post Natal Depression | 6 weeks following child birth
  Edinburgh Postnatal depression Scale

SECONDARY OUTCOMES:
General well being | 6 weeks following child birth
  General Physical and psychological well being was assessed using General Health Questionnaire
Parent-Infant Relationship | 6 weeks following child birth
  Parent-Infant Relationship Global Assessment Scale
Maternal Confidence | 6 weeks following child birth
  Maternal Self-Confidence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhari, Study Chair — Mothers Touch Foundation, India; Neha Sharma, Principal Investigator — Warwick Research Services; Sangram Birje, Study Director — Mothers Touch Foundation, India; Aparna Chaudhari, Study Director — Mothers Touch Foundation, India
Locations (1):
- NMP Medical Reserach Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided